CLINICAL TRIAL: NCT04359550
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter，Phase III Clinical Study of Recombinant Anti-PD-L1 Monoclonal Antibody (ZKAB001) for Maintenance Therapy in Patients With High-grade Osteosarcoma After Adjuvant Chemotherapy
Brief Title: Study of ZKAB001 for Maintenance Therapy in Patients With High-grade Osteosarcoma After Adjuvant Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NTL-LEES-2019-08
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: High-grade Osteosarcoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): ZKAB001 injection 10mg/kg once every 3 weeks for 1 cycle (Q3w), up to 16 cycles or 1 year of treatment.
  Interventions: Biological: Recombinant human anti-PD-L1 monoclonal antibody (ZKAB001)
- control group (Placebo Comparator): placebo will given in the same way for once every 3 weeks for 1 cycle (Q3w), up to 16 cycles or 1 year of treatment.
  Interventions: Other: placebo

INTERVENTIONS:
Biological: Recombinant human anti-PD-L1 monoclonal antibody (ZKAB001) — Recombinant human anti-PD-L1 monoclonal antibody (ZKAB001)
  Arms: treatment group
Other: placebo — placebo
  Arms: control group

SUMMARY:
It is a randomized, double-blind, placebo-controlled, multicenter study with the sample size is 362. The patients with high-grade osteosarcoma who had previously received surgery and completed adjuvant chemotherapy will be randomly assigned to ZKAB001 group (trial group) or placebo group (control group) according to 1:1. The purpose is to evaluate the efficacy and safety of ZKAB001 in maintenance therapy after adjuvant chemotherapy in patients with high-grade osteosarcoma.

DETAILED DESCRIPTION:
The patients will be given ZKAB001 injection in 10mg/kg or placebo once every 3 weeks for a total of 16 cycles or 1 year. The end point is that the patient has been taking the drug for 16 cycles or 1 year, or the patient dies or develops intolerable toxicity or confirmed disease recurrence or distant metastasis or withdrawal of informed consent, whichever comes first.

In this study, after a screening period of no more than 28 days, qualified subjects will be given ZKAB001 or placebo and test visits. Imaging examination will be performed every 12 weeks after the first dose until the local or distant recurrence of the disease, or the initiation of other systematic anti-tumor therapy or death, whichever come first.

The survival follow-up period starts from the last treatment to a maximum of 4 years, or to the death or loss of follow-up or withdrawal of informed consent or the sponsor terminates the study every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the trial and sign the informed consent form.
* Age ≥ 12 years old, both male and female.
* High-grade osteosarcoma diagnosed by histopathology (Ennecking stage II) ,radical surgery (R0 resection) and the adjuvant chemotherapy was confirmed by investigators. The end of adjuvant chemotherapy was no more than 12 weeks.
* Chemotherapy with more than two drugs must be used; the accumulated dose of doxorubicin should not be less than 300mg/m^2 (including converted dose); the total course of chemotherapy before and after operation should not be less than 12 times, the starting time of postoperative chemotherapy should not exceed 30 days, and the time of postoperative chemotherapy should not exceed 40 weeks.
* The score of the Eastern Cooperative Oncology Group (ECOG) is 0-1.
* The estimated survival time is more than 3 months.
* The functions of important organs meet the following requirements;

  1. Absolute neutrophil count ≥ 1.5 × 10^9 / L.
  2. Platelet count ≥ 75 × 10^9 /L.
  3. Hemoglobin ≥ 90g/L.
  4. Serum albumin ≥ 28g/L.
  5. Total bilirubin ≤ 1.5 × ULN;ALT, AST ≤ 2.5 × ULN.
  6. Serum creatinine ≤ 1.25 × ULN or endogenous creatinine clearance ≥ 50mL/min (using standard Crockcroft-Gault formula).
  7. Thyroid function: thyroid stimulating hormone (TSH) is normal. If TSH is abnormal, free thyroxine（ FT3 and FT4 ）levels should be examined. Normal FT3 and FT4 levels can be enrolled.
* Female subjects of childbearing age should take effective contraceptive methods during the study period and within 3 months after the end of the study period, and the serum human chorionic gonadotropin pregnancy test (HCG) must be negative within 7 days before enrollment.

Exclusion Criteria:

* Local recurrence or distant metastasis;
* There is active autoimmune disease or history of autoimmune disease (such as, but not limited to, interstitial pneumonia, uveitis, colitis, hepatitis, arthritis, glomerulonephritis, hypophysitis, hyperthyroidism, hypothyroidism, etc.), but does not include autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormones.
* Type I diabetes with stable doses of insulin;
* Vitiligo or cured childhood asthma / allergies in adults without medical intervention.
* The subjects were treated with immunosuppressants, or systemic or absorbable local corticosteroids with the purpose of immunosuppression (prednisone or equivalent for more than 10mg/ days), and continued to use them within 2 weeks before enrollment.
* Have received any form of organ transplantation, including allogeneic stem cell transplantation;
* Previously known to be allergic to macromolecular protein preparations or to any ZKAB001 components;
* Previous or simultaneous suffering from other malignant tumors (except those that have been cured or cancer-free for more than 5 years, such as basal cell carcinoma of the skin, carcinoma in situ of the cervix and papillary carcinoma of the thyroid, etc.);
* Uncontrolled cardiac clinical symptoms or diseases, such as heart failure above New York Heart Association(NYHA) 2, unstable angina pectoris, myocardial infarction within 1 year, clinical supraventricular or ventricular arrhythmias requiring intervention, echocardiography shows that the left ventricular ejection fraction at rest is less than 50%; - The completion of the treatment of radiotherapy, chemotherapy, surgery and/or molecular targeted therapy is less than 3 weeks before the first dose of study drug;
* Active infection (need to be treated with anti-bacterial, viral and/or fungal drugs), or fever of unknown origin occurred during the screening period and occurred within one week before the first dose (judged by the investigators, except the fever caused by tumor).
* Positive for human immunodeficiency virus (HIV); untreated active hepatitis B (hepatitis B surface antigen is positive and peripheral blood HBV-DNA titer ≥ 1000IU/ml or comply with local positive criteria) and/or hepatitis C (hepatitis C antibody is positive and HCV-RNA is higher than the lower limit)
* Patients with active pulmonary tuberculosis infection found by medical history or CT examination, or patients with active pulmonary tuberculosis infection within one year before entering the group, or patients with active pulmonary tuberculosis infection history more than one year ago but without formal treatment;
* Participating in other clinical studies, or less than 4 weeks from the end of the previous clinical study;
* Other systemic anti-tumor therapy may be received during the study period;
* Previously received other PD-1 and / or PD-L1, or CTLA-4 antibody therapy, or other drug therapy for immune receptor modulators;
* The live vaccine was vaccinated within 4 weeks before screening.
* Known history of psychotropic substance abuse, alcohol abuse or drug use;
* Pregnant or lactating women;
* Any mental state that hinders the understanding or provision of informed consent;
* The investigators consider that the patient had other factors that might lead to the termination of the study, such as other serious diseases or serious laboratory abnormalities or accompanied by other factors that would affect the safety of the subjects, or family or social factors that would affect the collection of data and samples.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
One-year DFS rate | 1 year
  The percentage of patients with no recurrence or metastasis within one year

SECONDARY OUTCOMES:
Five-years OS rate | 5 years
  Patients who survive within 5 years after the first dose.
adverse events | 5 years
  Incidence and severity of adverse events
Immunogenecity of ZKAB001 | 1 year
  To evaluated the number of subjects presenting detectable anti drug antibodies (ADAs).
PD-L1 expression | 1 year
  Correlation between PD-L1 expression level and clinical efficacy